CLINICAL TRIAL: NCT04331106
Title: Online-based Survey of the Anxiety Associated With the COVID-19 Pandemic in the General Population in Germany
Brief Title: Survey of the Anxiety Associated With the COVID-19 Pandemic
Acronym: CORA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Antonia Bendau, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: EA1/071/20
Record Dates: First submitted 2020-03-27; First posted 2020-04-02 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Anxiety Related to the COVID-19 Pandemic
Keywords: Anxiety; Pandemic; Corona-Virus; SARS-CoV-2; Corona; Covid-19; Public Health; Mental Health; Health; Mental Disorders
MeSH Terms: conditions — Anxiety Disorders; COVID-19; Psychological Well-Being; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Population in Germany: Reasonably large and representative sample of the general population in Germany
  Interventions: Diagnostic Test: Online Questionnaire

INTERVENTIONS:
Diagnostic Test: Online Questionnaire — Online Questionnaire via SoSci Survey

SUMMARY:
The study aims to systematically examine various aspects of the anxiety associated with the COVID-19 pandemic in Germany. The data collection is carried out online with longitudinal repeated measurements.

DETAILED DESCRIPTION:
The COVID-19 pandemic is currently one of the greatest challenges for numerous countries - also for Germany. In addition to its somatic and economic consequences, the psychological dimension of the Coronavirus pandemic is discussed increasingly and is visible in public life - e.g. in the "pandemic-caused experience of threat", "loss of control" and "panic" of multiple people. The study examines the phenomenon of this "corona-related anxiety" in terms of epidemiological, clinical and psychosocial characteristics. It is investigated how "corona anxiety" affects people who already have an anxiety disorder or other mental illnesses as well as formerly mentally healthy people. It is also examined how media reporting and personal consequences of COVID-19 are connected with corona-related anxiety and if there is a need for therapeutic support regarding corona-related anxiety.

To answer these questions a longitudinal online survey targeting the general population in Germany is carried out. The survey takes place all three weeks as long as the pandemic lasts and ends with one follow-up one year later.

ELIGIBILITY:
Inclusion Criteria:

* informed consent was given
* age ≥ 18
* able to complete the questionnaire in German
* country of residence: Germany

Exclusion Criteria:

* if at least one of the inclusion criteria is not met

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population in Germany
Sampling Method: Probability Sample
Enrollment: 7500 (Estimated)
Dates: Start 2020-03-27 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Characteristics of COVID-19-related anxiety | 1 day
  To investigate specific fears regarding the COVID-19 pandemic 9 self created items are used. Values ranging from 1 to 6, higher scores indicate a worse outcome.
COVID-19-related anxiety symptoms | 1 day
  Modified German version of the DSM-5 Severity-Measure-For-Specific-Phobia-Adult-Scale by Beesdo-Baum et al. (2014). 10 items, values ranging from 1 to 5, higher scores indicate a worse outcome. The Scale was adapted to anxiety symptoms related to COVID-19.

SECONDARY OUTCOMES:
Self-efficacy and coping with COVID-19 | baseline (1 day) + after 3 weeks + after 6 weeks + after 9 weeks + after 6 months + after 7 months + after 9 months + after 12 months
  Self-efficacy and coping with the COVID-19 pandemic are measured with 13 self created items. Values ranging from 1 to 6; higher scores indicate a better outcome (except inverted items).
Consequences of COVID-19 in the last three weeks. | baseline (1 day) + after 3 weeks + after 6 weeks + after 9 weeks + after 6 months + after 7 months + after 9 months + after 12 months
  Personal consequences of the COVID-19 pandemic in the last three weeks are collected with five self-created items.
General Illness Attitude | baseline (1 day) + after 3 weeks + after 6 weeks + after 9 weeks + after 6 months + after 7 months + after 9 months + after 12 months
  General illness attitudes are measured with 3 subscales (Worry about illness; Thanatophobia; Bodily preoccupations) of the German version of the Illness Attitude Scales (IAS) by Hiller & Rief (2004). 9 Items; values ranging from 1 to 5, higher scores indicate a worse outcome.
Media reporting | baseline (1 day) + after 3 weeks + after 6 weeks + after 9 weeks + after 6 months + after 7 months + after 9 months + after 12 months
  Frequency, effects and formats of consumed media related to COVID-19 are measured with 5 self created items.
Ultra-brief screening scale for anxiety and depression | baseline (1 day) + after 3 weeks + after 6 weeks + after 9 weeks + after 6 months + after 7 months + after 9 months + after 12 months
  To screen for general anxiety and depressive symptoms the German version of the Patient Health Questionnaire-4 (PHQ-4) by Löwe (2015) is used. 4 items; values ranging from 0 to 3, higher scores indicate a worse outcome.
Change in characteristics of COVID-19-related anxiety | baseline (1 day) + after 3 weeks + after 6 weeks + after 9 weeks + after 6 months + after 7 months + after 9 months + after 12 months
  To investigate specific fears regarding the COVID-19 pandemic 9 self created items are used. Values ranging from 1 to 6, higher scores indicate a worse outcome.
Change in COVID-19-related anxiety symptoms | baseline (1 day) + after 3 weeks + after 6 weeks + after 9 weeks + after 6 months + after 7 months + after 9 months + after 12 months
  Modified German version of the DSM-5 Severity-Measure-For-Specific-Phobia-Adult-Scale by Beesdo-Baum et al. (2014). 10 items, values ranging from 1 to 5, higher scores indicate a worse outcome. The Scale was adapted to anxiety symptoms related to COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Ströhle, Prof.Dr., Study Director — Charité-Universitätsmedizin Berlin - Department of Psychiatry and Psychotherapy; Antonia Bendau, M.Sc.Psych., Principal Investigator — Charité-Universitätsmedizin Berlin - Department of Psychiatry and Psychotherapy
Locations (1):
- Charité-Universitätsmedizin Berlin - Department of Psychiatry and Psychotherapy, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bendau A, Petzold MB, Strohle A, Plag J. Viral Transmission? A Longitudinal Study of Media Use and Its Relation to Mental Strain During the First 2 Years of the COVID-19 Pandemic. Int J Behav Med. 2025 Apr;32(2):214-226. doi: 10.1007/s12529-024-10293-3. Epub 2024 May 20. PMID 38769221
- [Derived] Bendau A, Petzold MB, Plag J, Asselmann E, Strohle A. Illness anxiety predicts higher mental strain and vaccine willingness-A nine-wave longitudinal study during the first 1.5 years of the COVID-19 pandemic in Germany. Stress Health. 2023 Dec;39(5):1137-1147. doi: 10.1002/smi.3255. Epub 2023 May 9. PMID 37158010
- [Derived] Olsson A, Olsson M, Fedorowski A, Hagell P, Wictorin K. The Orthostatic Hypotension Questionnaire in Swedish tested in patients with parkinsonism. Brain Behav. 2020 Sep;10(9):e01746. doi: 10.1002/brb3.1746. Epub 2020 Jul 7. PMID 32633094